CLINICAL TRIAL: NCT04369157
Title: The Role of Zinc and Inflammation in Susceptibility to Post-operative Cognitive Dysfunction
Brief Title: Zinc and Post-Operative Cognitive Dysfunction
Status: Withdrawn | Type: Observational
Why Stopped: As a result of Covid-19, this study did not proceed.
Sponsor: University of Reading (Other)
Collaborators: Royal Berkshire NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Prof Claire Williams, Professor, University of Reading
Other Study IDs: RDG-006
Record Dates: First submitted 2020-01-23; First posted 2020-04-30 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Elective Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma or serum samples processed to remove DNA, to determine zinc status and POCD biomarkers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elective surgery group: Patients undergoing hip/knee replacements or colorectal surgery will be recruited and tested on 3 occasions: pre-op, post-op and at follow-up. POCD status will be determined at post-op and follow up. Cognitive function, zinc status, POCD biomarkers and inflammatory markers will be measured on all 3 occasions.
  Interventions: Procedure: Elective surgery

INTERVENTIONS:
Procedure: Elective surgery — Patients will be scheduled to undergo elective orthopaedic (knee/hip replacement) or colorectal surgery.

SUMMARY:
A decline in cognitive abilities following surgery (POCD: Post-Operative Cognitive Dysfunction) affects up to 47% of patients undergoing a surgical procedure. Risk factors include age, previous depression, alcohol and drug use, smoking, cognitive impairment as well as pre-operative biochemical and haematological abnormalities. Inflammation has been proposed as a potential cause, however, there is little empirical and clinical evidence in this area to determine aetiology or reduce risk of incidence.

Zinc is an important metal for brain function, with deficiency associated with poorer cognitive outcomes. In relation to POCD, biomarker studies have revealed that levels of a zinc-alpha-2-glycoprotein (AZGP1) were lower in patients with POCD. AZGP1 is a multifunctional glycoprotein implicated in cell adhesion, immune response, transmembrane transport and cellular proliferation. Microglia, the immune cells of the brain, are highly sensitive to changes in zinc which have been proposed to contribute to neurodegenerative disease as well as POCD. However, whilst animal studies looking at the effects of zinc on cognition have been promising, robust human trials are lacking.

This research aims to establish the role of zinc in POCD by determining associations between zinc status, inflammation, cognitive function, and biomarkers of POCD risk and incidence. This will be achieved by gathering clinical and cognitive data from a sample of older adults undergoing surgery. Blood samples will be taken pre and post-operatively to establish zinc status and plasma concentrations of biomarkers of POCD risk and incidence. Pre and post-operative cognitive assessments will also be conducted to measure memory and executive function. Incidence of POCD will be determined via neurological assessment according to diagnostic criteria.

Should associations between zinc status, POCD biomarkers, inflammation, cognitive performance and POCD incidence be established, not only would it lead to future work to investigate potential mechanisms of action as well as intervention studies looking to support zinc status, optimising early identification of individuals who may be at higher risk of developing POCD should lead to better patient outcomes.

DETAILED DESCRIPTION:
Healthy older adults under-going elective surgery (knee replacement, hip replacement or colorectal surgery) will be recruited via the Royal Berkshire Hospital. Participants will be aged 60 years and above, will have the capacity to give fully informed consent and will be undergoing elective orthopaedic or colorectal surgery.

Participation will involve testing on 3 occasions: 48hours-3 weeks prior to surgery (in the participant's home), 1-3 days post-surgery (in the Royal Berkshire Hospital) and approximately one month post-surgery (in the participant's home).

On each occasion, the Montreal Cognitive Assessment (MoCA) and Confusion Assessment Method (CAM) will be administered along with various cognitive tests measuring executive function (Trials A & B, Stroop, Letter memory task, verbal fluency) and memory (the episodic memory tests of free recall and recognition from the CERAD: Consortium to Establish a Registry for Alzheimer's Disease neuropsychological test battery), as well as completion of questionnaires to determine mood (the Hospital Anxiety and Depression Scale [HADS] and the Positive and Negative Affect Scale [PANAS]) and sleep quality (the Pittsburgh Sleep Quality Index). The cognitive testing should take approximately 30-40 minutes.

At the first session (pre-operation) only, dietary information will also be collected via a food frequency questionnaire, as well as measures of fluid and crystallised intelligence (the National Adult Reading Test and Block Design from the Wechsler Adult Intelligence Scale - Revised respectively).

In addition, at each visit, a blood sample (maximum volume of 9mL, less than one tablespoon) will be taken from the participants for analysis of zinc concentration and markers of POCD and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or over
* Able to provide fully informed consent
* Scheduled to undergo orthopaedic (knee/hip replacement) or colorectal surgery
* English as their primary language

Exclusion Criteria:

* Under 60 years of age
* Unable to provide fully informed consent
* English not their primary language
* Not electing to undergo any surgery or surgery that is not a knee or hip replacement, or colorectal surgery

Ages: 60 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults aged over 60 years scheduled to undergo elective orthopaedic or colorectal surgery at the Royal Berkshire Hospital
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Baseline zinc status as a predictor of POCD incidence 1-3 days post-operation | 1-3 days post operation
  Concentration of zinc in plasma/serum at baseline as a predictor for development of POCD 1-3 days post operation
Baseline zinc status as a predictor of POCD incidence at follow-up | One month post operation
  Concentration of zinc in plasma/serum at baseline as a predictor for development of POCD at follow-up
POCD risk biomarker as a predictor of POCD incidence 1-3 days post operation | 1-3 days post operation
  Concentration of POCD risk biomarker AZGP1 in plasma/serum at baseline as a predictor for development of POCD 1-3 days post operation
POCD risk biomarker as a predictor of POCD incidence at follow-up | One month post operation
  Concentration of POCD risk biomarker AZGP1 in plasma/serum at baseline as a predictor for development of POCD at follow-up
Baseline cognitive function (global Z score) as a predictor of POCD incidence 1- 3 days post operation | 1-3 days post operation
  Baseline cognitive function (global Z score) as a predictor for development of POCD 1-3 days post operation
Baseline cognitive function (global Z score) as a predictor of POCD incidence at follow-up | One month post operation
  Baseline cognitive function (global Z score) as a predictor for development of POCD at follow-up

SECONDARY OUTCOMES:
Baseline zinc status as a predictor of cognitive function (global Z score) 1-3 days | 1-3 days post operation
  Concentration of zinc in plasma/serum at baseline as a predictor of cognitive function (global Z score) 1-3 days post operation
Baseline zinc status as a predictor of cognitive function (global Z score) at follow-up | One month post operation
  Concentration of zinc in plasma/serum at baseline as a predictor of cognitive function at follow-up
Current zinc status and incidence of POCD 1-3 days post operation | 1-3 days post operation
  Correlation between concentration of zinc in serum/plasma 1-3 days post
Current zinc status and incidence of POCD at follow-up | One month post operation
  Correlation between concentration of zinc in serum/plasma at follow-up and POCD incidence at follow-up
Current zinc status and cognitive function (global Z score) 1-3 days post operation | 1-3 days post operation
  Correlation between concentration of zinc in serum/plasma 1-3 days post operation and cognitive function (global Z score) 1-3 days post-operation
Current zinc status and cognitive function (global Z score) at follow-up | One month post operation
  Correlation between concentration of zinc in serum/plasma at follow-up and cognitive function (global Z score) at follow-up
POCD risk biomarker AZGP1 at baseline as predictor of cognitive function (global Z score) 1-3 days post operation | 1-3 days post operation
  Concentration of AZGP1 in plasma/serum at baseline as a predictor of cognitive function (global Z score) 1-3 days post operation
POCD risk biomarker AZGP1 at baseline as predictor of cognitive function (global Z score) at follow-up | One month post operation
  Concentration of AZGP1 in plasma/serum at baseline as a predictor of cognitive function (global Z score) at follow-up
Correlation between POCD biomarkers (IL-6 and IL-2) 1-3 days post operation and POCD incidence 1-3 days post operation | 1-3 days post operation
  Correlation between the concentration of POCD biomarkers (IL-6 and IL-2) in plasma/serum 1-3 days post-operation and development of POCD 1-3 days post operation
Correlation between POCD biomarkers (IL-6 and IL-2) at follow-up and POCD incidence at follow-up | One month post operation
  Correlation between the concentration of POCD biomarkers (IL-6 and IL-2) in plasma/serum at follow-up and development of POCD at follow-up
Correlation between POCD biomarkers (IL-6 and IL-2) 1-3 days post operation and cognitive function (global Z score) 1-3 days post operation | 1-3 days post operation
  Correlation between the concentration of POCD biomarkers (IL-6 and IL-2) in plasma/serum 1-3 days post-operation and cognitive function (global Z score) 1-3 days post operation
Correlation between POCD biomarkers (IL-6 and IL-2) at follow-up and cognitive function (global Z score) at follow-up | One month post operation
  Correlation between the concentration of POCD biomarkers (IL-6 and IL-2) in plasma/serum at follow-up and cognitive function (global Z score) at follow-up
Mediating influence of POCD risk biomarker AZGP1 at baseline on a correlation between baseline zinc status and POCD incidence 1-3 days post operation | 1-3 days post operation
  Baseline concentration of POCD risk biomarker AZGP1 in serum/plasma as a mediator of a correlation between concentration of zinc in plasma/serum at baseline and POCD incidence 1-3 days post operation
Mediating influence of POCD risk biomarker AZGP1 at baseline on a correlation between baseline zinc status and POCD incidence at follow-up | One month post operation
  Baseline concentration of POCD risk biomarker AZGP1 in serum/plasma as a mediator of a correlation between concentration of zinc in plasma/serum at baseline and POCD incidence at follow-up
Mediating influence of POCD risk biomarker AZGP1 at baseline on a correlation between baseline zinc status and cognitive function (global Z score) 1-3 days post operation | 1-3 days post operation
  Baseline concentration of POCD risk biomarker AZGP1 in serum/plasma as a mediator of a correlation between concentration of zinc in plasma/serum at baseline and cognitive function (global Z score) 1-3 days post operation
Mediating influence of POCD risk biomarker AZGP1 at baseline on a correlation between baseline zinc status and cognitive function (global Z score) at follow-up | One month post operation
  Baseline concentration of POCD risk biomarker AZGP1 in serum/plasma as a mediator of a correlation between concentration of zinc in plasma/serum at baseline and cognitive function (global Z score) at follow-up
Mediating influence of POCD biomarkers (IL-6 and IL-2) on a correlation between zinc status and cognitive function (global Z score) 1-3 days post operation | 1-3 days post operation
  Concentration of POCD biomarkers (IL-6 and IL-2) in serum/plasma 1-3 days post operation as a mediator of a correlation between concentration of zinc in plasma/serum and cognitive function (global Z score) 1-3 days post operation
Mediating influence of POCD biomarkers (IL-6 and IL-2) on a correlation between zinc status and cognitive function (global Z score) at follow-up | One month post operation
  Concentration of POCD biomarkers (IL-6 and IL-2) in serum/plasma at follow-up as a mediator of a correlation between concentration of zinc in plasma/serum and cognitive function (global Z score) at follow-up
Mediating influence of baseline mood (PANAS) on a correlation between baseline cognitive function (global Z score) and POCD incidence 1-3 days post operation | 1-3 days post operation
  Baseline mood (PANAS) as a mediator of a correlation between baseline cognitive function (global Z score) and POCD incidence 1-3 days post operation
Mediating influence of mood (PANAS) 1-3 days post operation on a correlation between baseline zinc status and cognitive function (global Z score) 1-3 days post operation | 1-3 days post operation
  Mood 1-3 days post operation (PANAS) as a mediator of a correlation between serum/plasma concentration of zinc at baseline and cognitive function (global Z score) 1-3 days post operation
Mediating influence of mood (PANAS) at follow-up on a correlation between baseline zinc status and cognitive function (global Z score) at follow-up | One month post operation
  Mood (PANAS) at follow-up as a mediator of a correlation between concentration of zinc in plasma/serum at baseline and cognitive function (global Z score) at follow-up
Mediating influence of mood (PANAS) at follow up on a correlation between zinc status and cognitive function (global Z score) at follow-up | One month post operation
  Mood (PANAS) at follow up as a mediator of a correlation between concentration of zinc in plasma/serum and cognitive function (global Z score) at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Claire Williams, PhD, Principal Investigator — University of Reading
Locations (2):
- United Kingdom (2):
  - School of Psychology and Clinical Languages, University of Reading, Reading, Berkshire
  - Royal Berkshire Hospital, Reading, Berkshrie

IPD SHARING:
Plan to Share IPD: Yes
Only anonymised data will be shared if requested.
Time Frame: Data will be available on request following publication of the findings.
Access Criteria: Data will be shared at the discretion of the Principle Investigator.